CLINICAL TRIAL: NCT01851850
Title: Continue Providing Care for Patient Who Participated in the BIA 9-1067-302 Clinical Trial
Brief Title: Continuation Treatment Protocol for Patient Who Participated in the BIA 9-1067-302 Clinical Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIA-91067
Record Dates: First submitted 2013-05-01; First posted 2013-05-13 (Estimated); Last update posted 2020-03-16 (Actual); Status verified 2013-01

CONDITIONS: Parkinson Disease
Keywords: PD; Off periods; quality of life; dyskinesia; end-off-dose motor fluctuations
MeSH Terms: conditions — Parkinson Disease; Dyskinesias | interventions — opicapone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Drug (Experimental)
  Interventions: Drug: Opicapone

INTERVENTIONS:
Drug: Opicapone — 25mg or 50mg once per day

SUMMARY:
The purpose of the study is to extend the use of opicapone 25 or 50mg once per day by subjects who participated in the BIA 9-1067-302 clinical trial according form 4a for additional three years.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis with PD
* subjects who are willing to participate in the trial.
* subjects who participated in the BIA 9-1067-302 clinical trial.

Exclusion Criteria:

* subjects who didn't take part at the BIA 9-1067-302 clinical trial.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-05; Primary Completion 2016-05-24 (Actual); Study Completion 2016-05-24 (Actual)

PRIMARY OUTCOMES:
off periods | 6 month
  number of "off" periods during the day without worsening dyskinesia.

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medical Center, Petach Tiqva, Central District, Israel

IPD SHARING:
Plan to Share IPD: No